CLINICAL TRIAL: NCT02602808
Title: Study of Peripheral Blood Non-coding RNAs as Diagnosis and Prognosis Biomarker for Acute Pancreatitis
Acronym: NCRNAP
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of gastroenterology department, Changhai Hospital
Other Study IDs: Pancreatitis Markers
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis; non-coding RNA; biological markers; receiver operating characteristic curve; post-ERCP pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples were collected from patients within the first 24 h after hospital admission. Also, blood samples were collected from patients at the time point of 24 hr after ERCP procedure. Serum, plasma and blood cells was isolated after blood collection by centrifugation at room temperature.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Severe acute pancreatitis group: Severe acute pancreatitis is characterised by persistent organ failure.
- Moderately severe acute pancreatitis: Moderately severe acute pancreatitis is characterised by the presence of transient organ failure or local or systemic complications in the absence of persistent organ failure.
- Mild acute pancreatitis: Mild acute pancreatitis is characterised by the absence of organ failure and the absence of local or systemic complications.
- post-ERCP pancreatitis: Patients with new onset of epigastric pain, an increase in pancreatic enzymes of at least three times the upper limit of the normal range within 24 hours after ERCP, and hospitalization for at least 2 nights.

SUMMARY:
It is important to identify patients with acute pancreatitis who are at risk for developing persistent organ failure early in the course of disease. The investigators evaluated whether peripheral blood non-coding RNAs, including microRNAs and long noncoding RNA (lncRNA), could serve as a good marker for detection of acute pancreatitis with persistent organ failure at early phase.

DETAILED DESCRIPTION:
Acute pancreatitis is a sudden inflammation of the pancreas. It can have severe complications and high mortality despite treatment. While mild cases are often successfully treated with conservative measures, such as fasting and aggressive intravenous fluid rehydration, severe cases may require admission to the intensive care unit or even surgery to deal with complications of the disease process. The diagnosis of severe acute pancreatitis at an early phase remain a major challenge for clinicians.

Therefore, many biologic markers have been studied in an effort to improve the diagnostic rate and determine the severity of acute pancreatitis but with disappointing results. Non-coding RNAs, including microRNAs and long noncoding RNA (lncRNA), have recently been validated to stably exist in peripheral blood. Several publications showed that it may serve as potential markers for various diseases, including cancer and inflammation. Our current study evaluated whether and which kind of non-coding RNAs could serve as good markers for severe acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who was diagnosed acute pancreatitis
* Male or female
* 18 Years and older
* written informed consent

Exclusion Criteria:

* Symptoms of acute pancreatitis present for more than 72 hours
* Age under 18 years
* Pregnancy
* patients unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 18 years of age or older who were hospitalized in our hospital with acute pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 1097 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
The level of non-coding RNAs in peripheral blood | At admission
  RNA quantification after extraction using RT-PCR

SECONDARY OUTCOMES:
serum urea nitrogen | At admission
  serum urea nitrogen quantification
serum creatinine | At admission
  serum creatinine quantification
APACHE II score at admission | At admission
  APACHE II score determined by Temperature, MAP, heart rate, respiratory rate, Pao2, arterial pH, HCO3, sodium, potassium, creatinine, hematocrit, WBC, Glasgow Coma Score, age, chronic health points
BISAP score at admission | At admission
  BISAP socre determined by BUN (>25 mg/dL), impaired mental status (Glasgow Coma Score <15), SIRS (≥2), age (>60 y), pleural effusion

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital
Locations (3):
- China (3):
  - Linyi People's Hospital, Linyi, Shandong
  - Changhai Hospital, Second Military Medical University, Shanghai
  - Department of Gastroenterology, Shanghai First People's Hospital, Shanghai

REFERENCES:
- [Derived] Zhu H, Zhou X, Sun X, Fu C, Li G, Dong X, Kong X, Su X, Du Y. Serum Exosomal miR-216a Contributes to Acute Pancreatitis-Associated Acute Lung Injury by Enhancing Endothelial Cell Vascular Permeability Through Downregulating LAMC1. Pancreas. 2025 Jul 1;54(6):e537-e546. doi: 10.1097/MPA.0000000000002467. PMID 39937877
- [Derived] Li L, Zhang Q, Feng Y, Kong F, Sun F, Xie P, Zhao J, Yu H, Zhou J, Wu S, Zhao S, Li Z, Liu F, Du Y, Kong X. A Novel Serum Exosomal MicroRNA Signature in the Early Prediction of Persistent Organ Failure in Patients With Acute Pancreatitis. Ann Surg. 2025 Jul 1;282(1):93-99. doi: 10.1097/SLA.0000000000006229. Epub 2024 Feb 7. PMID 38323410